CLINICAL TRIAL: NCT04258410
Title: Quercetin for Cardio-Skeletal Muscle Health and Estrogen Deficiency (QUICKENED) Feasibility Study in Older Women
Brief Title: Quercetin for Cardio-Skeletal Muscle Health and Estrogen Deficiency
Acronym: QUICKENED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Per PI: "Never went to IRB Never recruited anyone Never resubmitted the score NIH application I am leaving the institution"
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-PENDING-LG
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Menopause Related Conditions
Keywords: estrogen deficiency; post-menopause; cardiac diastolic function; skeletal muscle function; skeletal muscle structure; cardiac structure
MeSH Terms: interventions — Quercetin; Flavonoids

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled parallel pilot trial of Quercetin vs placebo oral administration in 24 postmenopausal women.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled participants who complete the pre-treatment assessment will be randomly assigned to Quercetin or placebo. The trial manager who is not involved in any outcome assessments will carry out randomization following the protocol designed by the study biostatistician (Dr. Leng) prior to the study's start. The randomization sequence list will remain concealed from the investigators. Participants will be randomized using a computer-generated, password-protected randomization list, and simple randomization scheme. All staff involved in data collection and management will be kept unaware of the participants' group assignments and will explicitly inform participants that they (staff) are to remain blinded during the course of the study. The biostatistician will also be unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Blinded subjects in this arm will receive 2 placebo (blank) soft chews, twice daily, orally for 20 weeks.
  Interventions: Drug: Placebo oral soft chew
- Active Drug (Experimental): Blinded subjects in this arm will receive 1 g/day of Quercetin delivered in 2 soft chews (250 mg/chew), twice daily, orally, for 20 weeks.
  Interventions: Drug: Quercetin

INTERVENTIONS:
Drug: Placebo oral soft chew — placebo identical to experimental drug contained in soft chew
  Arms: Placebo
Drug: Quercetin — experimental drug contained in soft chew
  Other Names: Bioflavonoid
  Arms: Active Drug

SUMMARY:
Double blind randomized controlled parallel pilot trial of Quercetin vs placebo oral administration in 24 postmenopausal women. The study team will conduct a feasibility pilot in preparation for a larger efficacy trial that will test the protective effects of quercetin against cardiac and skeletal muscle dysfunction and changes in structure induced by estrogen loss and potential mechanistic pathways in post-menopausal women at risk of heart failure with preserved ejection fraction (HFPEF).

DETAILED DESCRIPTION:
Participants receive either oral Quercetin 1000 g/day or placebo for 20 weeks. Quercetin levels, biomarkers, ultrasounds (heart and muscle), functional assessments will be measured on enrollment and after the intervention. The study coordinator will contact participants weekly to monitor safety and ensure compliance. All quercetin administration will be supervised by Claudia L Campos, MD, Associate Professor of Internal Medicine, Medical Director Internal Medicine clinic.

ELIGIBILITY:
Inclusion Criteria:

* Female, postmenopausal, aged 60 to 74
* Stated willingness to comply with all study procedures and availability for the duration of the study
* High risk of Heart failure with preserved ejection fraction (HFPEF) using web-based Primary Care Physician-HF risk tool (Khan S, et al.10-Year Risk Equations for Incident Heart Failure in the General Population. Information used for calculation include: age, gender, race, hypertension treatment (yes or no), fasting glucose value, smoking status, body mass index, systolic BP, diabetes treatment (yes or no), total cholesterol, HDL cholesterol, and electrocardiogram QRS duration. Prospective participant's with scores >= 10% will be included.
* Electrocardiogram (EKG) on medical record

Exclusion Criteria:

* History of congestive heart failure or use of loop diuretics
* Recent myocardial infarction (MI), stroke, angina, or atrial fibrillation (in the past 6 months), either self-reported and or in the electronic medical record.
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Significant renal insufficiency requiring dialysis or estimated glomerular filtration rate (eGFR) < 15 mL/min
* Liver disease
* Psychiatric disease - uncontrolled major psychoses, depressions, dementia, or personality disorder
* Participants reporting extreme energy intakes >3500 or <500 kcal/day
* Plans to leave area within the study period
* Refuses informed consent

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Number of enrolled participants per month | up through 13 months
  Proportion of eligible participants enrolled each month, over the course of recruitment.
Eligibility: Proportion eligible after screening | baseline
  Proportion of eligible participants that are invited to participate after initial screening and reasons for declining enrollment.

SECONDARY OUTCOMES:
Adherence: Percent adherence to study visits | 20 weeks
  Missing data will be quantified, and reasons for failure to follow-up will be determined through informal comments from participants, via phone contact, to assess adherence barriers.
Adherence: Percent adherence to intervention | 20 weeks
  Participant treatment compliance will be determined by average plasma quercetin levels, in mg/dL, in each group.
Retention: Number of Subjects Lost to Follow Up | 20 weeks
  Missing data and drop-out will be quantified, and reasons for lost to follow up will be evaluated through informal comments from participants and Likert-ranked questions to assess participant perceptions of strengths and weaknesses of the study.
Retention: Number of Subjects Discontinued | 20 weeks
  Participants that are prematurely terminated or discontinued from the study will be quantified. The circumstances that may warrant discontinuation will be evaluated and recorded.
Acceptability: Changes in patient satisfaction | Baseline and week 20
  Likert-ranking to assess participant perceptions of the strengths and weaknesses of the study. Scores range from 1 to 5 with a higher score denoting a positive outcome.

OTHER OUTCOMES:
Changes in left ventricular systolic function | Baseline and 20 weeks
  Measure left ventricular ejection fraction (LVEF) by transthoracic echocardiogram (TTE), pre and post intervention
Changes in left ventricular diastolic function | Baseline and 20 weeks
  Measures of myocardial relaxation by early septal mitral annular velocity (e') via tissue Doppler, and early-to-late transmitral filling velocity ratios (E/A) via Doppler from transthoracic echocardiogram, pre and post intervention
Changes in left ventricular filling pressure | Baseline and 20 weeks
  Calculate ratio of early transmitral filling (E)-to-mitral annular velocity (e'), or E/e', by Doppler-derived images from TTE, pre and post intervention
Changes in left ventricular (LV) structure | Baseline and 20 weeks
  Calculate LV mass and relative wall thickness from standard TTE images, pre and post intervention
Changes in left atrial structure | Baseline and 20 weeks
  Measure left atrial volume by TTE, pre and post intervention
Changes in skeletal muscle quality | Baseline and 20 weeks
  Echo-intensity, in pixels, of the vastus lateralis muscle of the thigh will be measured using ultrasound, pre and post intervention.
Changes in skeletal muscle composition | Baseline and 20 weeks
  Measure subcutaneous fat adjacent to vastus lateralis muscle by ultrasound, pre and post intervention
Changes in exercise capacity | Baseline and 20 weeks
  6-minute walk distance (6 MWD), pre and post intervention
Changes in skeletal muscle strength | Baseline and 20 weeks
  Five times sit-to-stand test, pre and post intervention
Changes in biomarker of inflammation | Baseline and 20 weeks
  Blood sample for measure of high-sensitivity C-reactive protein (hs-CRP), pre and post intervention
Changes in biomarker of oxidative stress | Baseline and 20 weeks
  Blood sample for determination of malondialdehyde by ELISA assay, pre and post intervention
Changes in biomarker of anti-oxidant defense | Baseline and 20 weeks
  Blood sample for glutathione levels using a commercial assay kit, pre and post intervention
Changes in biomarker of LV remodeling | Baseline and 20 weeks
  Blood sample for N terminal-ProBNP levels using the Roche Assay, pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Groban, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No